CLINICAL TRIAL: NCT04880850
Title: A 26-week Trial Comparing the Effect and Safety of Once Weekly Insulin Icodec and Once Daily Insulin Glargine 100 Units/mL, Both in Combination With Bolus Insulin With or Without Non-insulin Anti-diabetic Drugs, in Subjects With Type 2 Diabetes on a Basal-bolus Regimen
Brief Title: A Research Study to Compare Two Types of Insulin, a New Weekly Insulin, Insulin Icodec and an Available Daily Insulin, Insulin Glargine, Both in Combination With Mealtime Insulin, in People With Type 2 Diabetes Who Use Daily Insulin and Mealtime Insulin (ONWARDS 4)
Acronym: ONWARDS 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4480; U1111-1247-5269 (Other: World Health Organization (WHO)); 2020-000474-16 (EudraCT Number)
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- insulin icodec + insulin aspart (Experimental): Participants will get once weekly injections in combination with 2-4 times daily injections of insulin aspart
  Interventions: Drug: Insulin icodec; Drug: Insulin aspart
- Insulin glargine + insulin aspart (Active Comparator): Participants will get once daily injections in combination with 2-4 times daily injections of insulin aspart
  Interventions: Drug: Insulin glargine; Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin icodec — Participants will receive subcutaneous (s.c.) injections of insulin icodec once weekly for 26 weeks
  Arms: insulin icodec + insulin aspart
Drug: Insulin glargine — Participants will receive subcutaneous (s.c.) injections of insulin glargine once daily for 26 weeks
  Arms: Insulin glargine + insulin aspart
Drug: Insulin aspart — Participants will receive subcutaneous (s.c.) injections of insulin aspart 2-4 times daily for 26 weeks

SUMMARY:
This study compares insulin icodec (a new insulin taken once a week) to insulin glargine (an insulin taken once daily which is already available on the market) in people with type 2 diabetes.

The study will look at how well insulin icodec taken weekly controls blood sugar compared to insulin glargine taken daily.

Participants will either get insulin icodec that participants will have to inject once a week on the same day of the week or insulin glargine that participants will have to inject once a day at the same time every day. Which treatment participants will get is decided by chance. Participants will also get a mealtime insulin.The insulin is injected with a needle in a skin fold in the thigh, upper arm or stomach.

The study will last for about 8 months. participants will have 17 clinic visits and 13 phone calls with the study doctor.At 8 clinic visits participants will have blood samples taken. At 4 clinic visits participants cannot eat or drink (except for water) for 8 hours before the visit. Participants will be asked to wear a sensor that measures their blood sugar all the time in 3 periods for a total of 13 weeks (about 3 months) during the study.

Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged above or equal to 18 years at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus (T2D) greater than or equal to 180 days prior to the day of screening.
* Glycated haemoglobin (HbA1c) from 7.0-10.0% (53.0 85.8 mmol/mol) both inclusive at screening confirmed by central laboratory analysis.
* Treated with once daily basal insulin (neutral protamine hagedorn insulin, insulin degludec, insulin detemir, insulin glargine 100 units/mL, or insulin glargine 300 units/mL) and 2-4 daily injections of bolus insulin analog (insulin aspart, faster acting insulin aspart, insulin lispro, insulin glulisine) greater than or equal to 90 days prior to the day of screening with or without any of the following anti-diabetic drugs/regimens with stable doses greater than or equal to 90 days prior to screening:

Metformin / Sulfonylureas / Meglitinides (glinides) / DPP-4 inhibitors / SGLT2 inhibitors / Thiazolidinediones / Alpha-glucosidase inhibitors / Oral combination products (for the allowed individual oral anti-diabetic drugs) / Oral or injectable GLP-1-receptor agonists

* Body mass index (BMI) below or equal to 40.0 kg/m^2.

Exclusion Criteria:

* Any episodes (as declared by the subject or in the medical records.) of diabetic ketoacidosis within 90 days prior to the day of screening.
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening.
* Chronic heart failure classified as being in New York Heart Association Class IV at screening.
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or corticosteroids).
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (116):
- United States (52):
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - John Muir Physicians Network, Concord, California
  - Valley Research, Fresno, California
  - Diabetes/Lipid Mgmt & Res Ctr, Huntington Beach, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Clinical Trials Research_Sacramento_0, Sacramento, California
  - Diabetes Research Center, Tustin, California
  - Coastal Metabolic Research Center, Ventura, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Chase Medical Research LLC, Waterbury, Connecticut
  - MedStar Diabetes Institute, Washington D.C., District of Columbia
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - Clinical Trial Res Assoc,Inc, Plantation, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Physicians Research Assoc. LLC, Lawrenceville, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Saltzer Medical Group Research, Nampa, Idaho
  - Velocity Clin. Res Valparaiso, Valparaiso, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - MassResearch, LLC, Waltham, Massachusetts
  - Jefferson City Medical Group, PC, Jefferson City, Missouri
  - VA NEB - Western IA Health Stm, Omaha, Nebraska
  - Methodist Physicians Clin, Omaha, Nebraska
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - AMC Community Endocrinology, Albany, New York
  - Northport VA Medical Center_Northport_0, Northport, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Mountain Diabetes & Endocrine Center, Asheville, North Carolina
  - Physician's East Endocrinology, Greenville, North Carolina
  - Your Diabetes Endocrine Nutrition Group, Inc., Mentor, Ohio
  - Oregon Health & Science University_Portland_0, Portland, Oregon
  - Indiana-Armstrong Endocrinology Associates, Indiana, Pennsylvania
  - Prisma Health-Upstate, Greenville, South Carolina
  - AM Diabetes And Endocrinology Center, Bartlett, Tennessee
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Vanderbilt Diab Obes Clin Tri, Nashville, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Texas Diab & Endo, P.A., Austin, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Osvaldo A. Brusco MD PA, Corpus Christi, Texas
  - Baylr Sctt White Rs Inst, Endo, Dallas, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Protenium Clinical Research_Hurst, Fort Worth, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Capital Clin Res Ctr,LLC, Olympia, Washington
- Belgium (5):
  - Imeldaziekenhuis - Bonheiden - Department of Endocrinology, Bonheiden
  - CHU Helora - Site Warquignies, Boussu
  - Cliniques Universitaires Saint-Luc - Serv Endocrinologie - Diabétologie, Brussels
  - UZA - UZ Antwerpen - Department of Endocrinology, Edegem
  - UZ Leuven - Endocrinology, Leuven
- India (17):
  - Kurnool Medical Collage, Kurnool, Andhra Pradesh
  - Medanta - The Medicity Multi-Speciality Hospital, Gurugram, Gurgaon, Haryana
  - St.John's Hospital, Bangalore, Karnataka
  - Bangalore Clinisearch, Bangalore, Karnataka
  - Lifecare Hospital and Research Centre, Bangalore, Karnataka
  - Belgaum Diabetes Centre, Belagavi, Karnataka
  - Manipal Hospital, Hebbal, Bengaluru, Bengaluru, Karnataka
  - Renai Medicity, Kochi, Kerala
  - Prince Aly Khan Hospital, Mumbai, Maharashtra
  - BSES MG hospital, Mumbai, Maharashtra
  - Grant Medical Foundation, Pune, Maharashtra
  - Max Super Speciality Hospital, Saket, New Delhi, National Capital Territory of Delhi
  - Fortis Hospital, Shalimar Bagh, New Delhi, New Delhi, National Capital Territory of Delhi
  - Maulana Azad Medical College, Delhi, New Delhi
  - All India Institute of Medical Sciences, New Dehli, New Delhi
  - S.C.B. Medical College, Cuttack, Odisha
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
- Italy (6):
  - A.O.U. Università Studi della Campania "Luigi Vanvitelli", Napoli, Campania
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro, Cz
  - Istituto Scientifico San Raffaele, Milan, MI
  - A.O.Universitaria S.ORSOLA-MALPIGHI - U.O.Endocrinologia e Cura, Bologna
  - Università degli Studi G. D'Annunzio, Chieti
  - Universita Degli Studi Di Roma La Sapienza - Policlinico Umberto I Medicina Sperimentale, Roma
- Japan (9):
  - Hayashi Diabetes Clinic_Internal Medicine and Diabetes Medicine, Chigasaki-shi, Kanagawa, Japan
  - Futata Tetsuhiro Clinic Meinohama_Internal medicine, Fukuoka-shi, Fukuoka
  - Sasaki Internal Medicine, Hokkaido
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Sugimoto Clinic,Internal Medicine, Kitakyusyu-shi, Fukuoka
  - Shimizu Clinic Fusa, Saitama
  - Oyama East Clinic_Internal Medicine, Tochigi
  - The Jikei University Hospital Dept of Diabetes, Metabolic, Tokyo
  - Noritake Clinic, Ushiku-shi, Ibaraki
- Mexico (3):
  - Centro de Investigacion Medica de Occidente S.C., Zapopan, Jalisco
  - Hospital Universitario Dr. José Eleuterio González_Monterrey, Monterrey, Nuevo León
  - Unidad Biomedica Avanzada Monterrey, Monterrey, Nuevo León
- Netherlands (7):
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Maxima Medisch Centrum, Eindhoven
  - Bethesda Diabetes Research Center en Bethesda ziekenhuis, Hoogeveen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Ikazia Ziekenhuis, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Romania (6):
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest, Bucurestii
  - Spitalul Judetean de Urgenta Targoviste, Târgovişte, Dâmbovița County
  - Sc Mediab Srl, Târgu Mureş, Mureș County
  - Mariodiab Clinic SRL, Brasov
  - S.C. Medcon S.R.L, Buzău
  - Clinical Emergency Sf. Apostol Andrei Hospital, Galati
- Russia (11):
  - Tumen State Medical University, Tyumen, Russia
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - City Hospital #5, Barnaul
  - KSFMU, Inrereginal Clinical Diagnostic center, Kazan'
  - Kirov Clinical Hospital #7, Kirov
  - Limited Liability Company "AriVa-Med", Kursk
  - City Clinical Hospital №52, Moscow
  - LLC "Centr Targetnoy Terapii", Moscow
  - Limited Law Company "Healthy Family" Medicine Center", Novosibirsk
  - SPb SBHI City Outpatient clinic #37, Saint Petersburg
  - Regional clinical cardiology dispensary, Saratov

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Philis-Tsimikas A, Bajaj HS, Begtrup K, Cailleteau R, Gowda A, Lingvay I, Mathieu C, Russell-Jones D, Rosenstock J. Rationale and design of the phase 3a development programme (ONWARDS 1-6 trials) investigating once-weekly insulin icodec in diabetes. Diabetes Obes Metab. 2023 Feb;25(2):331-341. doi: 10.1111/dom.14871. Epub 2022 Oct 14. PMID 36106652
- [Result] Mathieu C, Asbjornsdottir B, Bajaj HS, Lane W, Matos ALSA, Murthy S, Stachlewska K, Rosenstock J. Switching to once-weekly insulin icodec versus once-daily insulin glargine U100 in individuals with basal-bolus insulin-treated type 2 diabetes (ONWARDS 4): a phase 3a, randomised, open-label, multicentre, treat-to-target, non-inferiority trial. Lancet. 2023 Jun 10;401(10392):1929-1940. doi: 10.1016/S0140-6736(23)00520-2. Epub 2023 May 5. PMID 37156252
- [Derived] Mohan V, Kesavadev J, Murthy LS, Anil G, Chandrappa M, Kar S, Mishra S. Efficacy and Safety of Once-Weekly Insulin Icodec in Indian Participants with Diabetes: Results from ONWARDS 1, 4, and 6 Studies. Diabetes Ther. 2025 Nov;16(11):2193-2212. doi: 10.1007/s13300-025-01799-4. Epub 2025 Oct 6. PMID 41051694
- [Derived] Philis-Tsimikas A, Krogsdahl Bache J, Fu A, Kellerer M, Salvesen-Sykes K, Bain SC. Insights on Hospitalisations from the Phase 3a ONWARDS 1-6 Trials of Once-Weekly Insulin Icodec. Diabetes Ther. 2025 Aug;16(8):1615-1631. doi: 10.1007/s13300-025-01745-4. Epub 2025 Jun 4. PMID 40465144
- [Derived] Riddell MC, Heller S, Carstensen L, Rocha TMP, Kehlet Watt S, Woo VC. The effect of once-weekly insulin icodec vs once-daily basal insulin on physical activity-attributed hypoglycaemia in type 2 diabetes: a post hoc analysis of ONWARDS 1-5. Diabetologia. 2025 Jul;68(7):1416-1422. doi: 10.1007/s00125-025-06414-6. Epub 2025 Apr 5. PMID 40186685
- [Derived] Watada H, Asbjornsdottir B, Nishida T, Nishimura R, Yamamoto Y, Yamauchi T, Kadowaki T. Efficacy and safety of once-weekly insulin icodec versus once-daily basal insulin in Japanese individuals with type 2 diabetes: A subgroup analysis of the ONWARDS 1, 2 and 4 trials. Diabetes Obes Metab. 2024 Dec;26(12):5882-5895. doi: 10.1111/dom.15960. Epub 2024 Sep 30. PMID 39344833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 83 sites in 9 countries as follows: Belgium (5), India (9), Italy (6), Japan (9), Mexico (3), Netherlands (5), Romania (6), Russia (10), United States (30).
Pre-assignment Details: The trial duration is approximately 33 weeks, consisting of a 2-week screening period, followed by a 26-week randomised treatment period and a 5-week follow-up period.
Groups:
- Insulin Icodec: Participants were to receive once weekly subcutaneous (s.c.) injection of Insulin icodec for 26 weeks, using PDS290 prefilled pen-injector in combination with insulin aspart at a starting dose of 7 times the pre-trial total daily basal insulin dose + 50% of their 7 times total daily basal insulin dose. The following weekly dose was 7 times the total daily dose of the respective participants ('unit to unit switch' approach: current daily dose x 7). Participants were to perform once daily pre-breakfast self-monitoring plasma glucose (SMPG). The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: lesser than (<) 4.4 millimoles per liter (mmol/L): dose reduced by 20 units (U); 4.4-7.2 mmol/L: no adjustment; greater than (>) 7.2 mmol/L: dose increased by 20 U. Dose titration of insulin aspart was based on the respective premeal(s) and bedtime SMPG measured.
- Insulin Glargine: Participants were to receive once daily s.c. injection of Insulin glargine for 26 weeks, using SoloSTAR pre-filled pen-injector in combination with insulin aspart. Participants were to perform daily SMPG. The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 mmol/L: dose reduced by 3 U; 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: dose increased by 3 U. Dose titration of insulin aspart was based on the respective premeal(s) and bedtime SMPG measured.
Period: Overall Study
Arm/Group | Insulin Icodec | Insulin Glargine
Started | 291 | 291
Full Analysis Set (FAS) | 291 | 291
Safety Analysis Set (SAS) | 291 | 291
Completed | 275 | 273
Not Completed | 16 | 18
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 3 | 6
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 9 | 10

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants from baseline (week 0) to week 26.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Icodec | Insulin Glargine | Total
Number analyzed (Participants) | 291 | 291 | 582
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.67 (10.13) | 59.91 (9.92) | 59.79 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 141 | 278
  Male | 154 | 150 | 304
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 53 | 105
  Not Hispanic or Latino | 239 | 237 | 476
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 95 | 93 | 188
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 13 | 8 | 21
  White | 183 | 187 | 370
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline (week 0) to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: Baseline (week 0), Week 26
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%) of HbA1c
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 291 | 291
Percentage (%) of HbA1c | -1.16 (0.05) | -1.18 (0.05)
Statistical Analysis 1: Comparison: Insulin Icodec vs Insulin Glargine; The response and change from baseline in response after 26 weeks were analysed using an analysis of covariance (ANCOVA) model with treatment, region and personal continuous glucose monitoring (CGM) device use as fixed factors, and baseline response as covariate; Test type: Non-Inferiority — Non-inferiority of insulin icodec was considered confirmed if the upper limit of the two-sided 95% confidence interval (CI) for mean treatment difference (insulin icodec minus insulin glargine) was strictly below 0.3%; p < 0.0001, ANCOVA; Treatment difference = 0.02, 95% CI 2-sided [-0.11 to 0.15]

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline (week 0) to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: Baseline (week 0), Week 26
Population: Full analysis set included all randomised participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 283 | 284
Millimoles per liter (mmol/L) | -1.75 (0.16) | -1.61 (0.16)

3. Secondary Outcome: Percentage of Time in Target-range 3.9-10.0 mmol/L (70-180 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time in target-range 3.9-10.0 mmol/L (70-180 milligrams per deciliter [mg/dL]) using continuous glucose monitoring (CGM) system from week 22 to week 26 is presented. Time in target range is defined as 100 times the number of recorded measurements in glycaemic target range 3.9-10.0 mmol/L (70-180 mg/dL), both inclusive, divided by the total number of recorded measurements. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: From week 22 to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage (%) of time
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 244 | 237
Percentage (%) of time | 66.88 (15.62) | 66.44 (16.17)

4. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. The outcome data was evaluated based on the on-treatment observation period. The on-treatment observation period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit, the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period.
Time Frame: From baseline (week 0) to week 31
Population: Safety analysis set included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 291 | 291
Episodes | 7 | 3

5. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL) Confirmed by Blood Glucose (BG) Meter)
Description: Clinically significant hypoglycaemic episodes (level 2) were defined as episodes that were sufficiently low to indicate serious, clinically important hypoglycaemia with plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL). The outcome data was evaluated based on the on-treatment observation period. The on-treatment observation period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit, the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period.
Time Frame: From baseline (week 0) to week 31
Population: as for outcome 4
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 291 | 291
Episodes | 937 | 935

6. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Clinically significant hypoglycaemic episodes (level 2) were defined as episodes that were sufficiently low to indicate serious, clinically important hypoglycaemia with plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL). Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. The outcome data was evaluated based on the in-trial observation period. The on-treatment observation period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit, the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period.
Time Frame: From baseline (week 0) to week 31
Population: as for outcome 4
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 291 | 291
Episodes | 944 | 938

7. Secondary Outcome: Percentage of Time Spent Below 3.0 mmol/L (54 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time spent less than (<) 3.0 mmol/L (54 mg/dL) using CGM system from week 22 to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: From week 22 to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage (%) of time
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 244 | 237
Percentage (%) of time | 0.73 (1.14) | 0.61 (1.07)

8. Secondary Outcome: Percentage of Time Spent Above 10 mmol/L (180 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time spent > 10 mmol/L (180 mg/dL) using CGM system from week 22 to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: From week 22 to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage (%) of time
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 244 | 237
Percentage (%) of time | 30.47 (15.90) | 31.30 (16.67)

9. Secondary Outcome: Mean Weekly Insulin Dose
Description: Estimated mean weekly insulin dose during the last 2 weeks of treatment (from week 24 to week 26) is presented. The outcome data was evaluated based on the on-treatment observation period. The on-treatment observation period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit, the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period.
Time Frame: From week 24 to week 26
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units of insulin
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 273 | 266
Units of insulin | 513.54 [486.10 to 542.52] | 559.05 [528.63 to 591.22]

10. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: Baseline (week 0), Week 26
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | Insulin Icodec | Insulin Glargine
Number analyzed (Participants) | 291 | 291
Kilograms (kg) | 2.73 (0.29) | 2.16 (0.40)

ADVERSE EVENTS:
Time Frame: From baseline (week 0) to week 31.
Description: All presented AEs are treatment emergent. Treatment emergent adverse events (TEAEs): events that had onset date during on-treatment period, time period in which participants was considered exposed to trial product. Safety analysis set included all randomised participants randomly assigned to trial treatment who took at least 1 dose of trial product.
Arm/Group | Insulin Icodec | Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 2/291 | 1/291
Serious Adverse Events (participants affected / at risk) | 22/291 | 25/291
Other Adverse Events (participants affected / at risk) | 48/291 | 44/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=291) | Insulin Glargine (N=291)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (3)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (3) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=291) | Insulin Glargine (N=291)
COVID-19 (Infections and infestations) | 25 (25) | 22 (24)
Diabetic retinopathy (Eye disorders) | 12 (14) | 15 (15)
Diarrhoea (Gastrointestinal disorders) | 15 (18) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT04880850/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04880850/SAP_001.pdf